CLINICAL TRIAL: NCT03227718
Title: VOR Suppression in Non-Gymnast Adults
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: HM20008030
Record Dates: First submitted 2017-06-08; First posted 2017-07-24 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Vestibular; Performance
Keywords: VOR
MeSH Terms: interventions — Reflex, Vestibulo-Ocular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- athletic background: ex-gymnasts
  Interventions: Behavioral: VOR and coordination measurements
- control: age-matched non-gymnastics background
  Interventions: Behavioral: VOR and coordination measurements

INTERVENTIONS:
Behavioral: VOR and coordination measurements — measurement of VOR and VOR suppression in addition to hand-eye coordination tasks

SUMMARY:
The researchers hypothesize that there is a correlation between Vestibulo-ocular reflex (VOR) performance and innate athletic skill level. A similar study was conducted in female, young adult gymnasts where a correlation was shown between VOR performance and gymnastic skill level. However, the results from this study did not suggest that VOR differences develop as a result of practice; rather that the differences in VOR may simply allow some individuals to become better performers. In this study the researchers would like to extend the population to adults both with and without a background in gymnastics to determine the natural relationship between VOR and innate athletic potential.

DETAILED DESCRIPTION:
Sports like gymnastics, diving, and ice skating often involve rotational elements with high angular velocities. Many of these are airborne skills and have a significant element of risk. The athletes who perform these skills have to rely on sensory information from the visual and vestibular systems. It has been suggested that the vestibular system adapts to these types of inputs and the athlete no longer experiences dizziness associated with multiple rotations.

A recent Neuroscience abstract described a small study of the directional selectivity of vestibular habituation adult professional figure skaters. The results showed that figure skaters demonstrated a profound reduction in the magnitude of post-rotary nystagmus and caloric test response in their preferred direction of rotation. It was suggested that this sensitivity was a result of "habituation." The authors implied that the skaters learned to suppress vestibular receptors on the side that they turned toward. This deduction is based on patients that develop pathology on one side and learn to suppress the sensation on that side. However, we do not currently know if the developing vestibular system works the same way or if this is an inherited trait. Most of these athletes started as children, when their vestibular system was still developing, and may have a more fine-tuned vestibular system and be able to suppress certain reflexes. On the other hand, it could be that some people are born with the ability to suppress this sensation, thus allowing them to become elite athletes. Currently there isn't a defined relationship between a person's athleticism or athletic upbringing and their vestibular system performance.

A major component of vestibular performance is the Vestibular Ocular Reflex (VOR). The VOR is responsible for stabilizing the visual field on the retina during head movement. To accomplish this, the eyes are reflexively moved in a direction opposite the head. For example, in a twisting gymnast, this actually reduces the ability of gymnasts to see the landing during airborne skills. Hence, it becomes necessary for gymnasts to cancel or suppress their VOR in order to view the landing. A previous study conducted by the researchers determined that young, actively practicing gymnasts (mean age 15±2.2) had a higher ability to suppress their VOR than non-gymnasts of the same age. This previous study determined that there is a correlation between VOR performance and gymnastic skill level. However, these results do not suggest that the VOR differences develop as a result of practice.

This study aims to establish a relationship between VOR performance and athleticism. By comparing ex-gymnast adults (ages 18-30), and their age-matched, non-gymnast counterparts to the previous study results involving actively practicing, child gymnasts, a relationship between VOR performance and athletic skill can be determined. Furthermore, examining the VOR data collected from this study to data collected from tests aimed at determining athleticism, or a person's athletic potential, it may be possible to relate VOR performance to athletic skill; In other words, determining whether athletes are successful because their vestibular performance is superior to those whom are non-athletes, or it is a learned skill with practice.

ELIGIBILITY:
Inclusion Criteria:

* Normal, adults will be recruited from the University community via a sample of convenience.

Exclusion Criteria:

* Children under the age of 18.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Approximately 12 adults (6 ex-gymnastics, and 6 age matched, non-gymnast counterparts), ages 18-30 will be obtained via a sample of convenience from the University community. Subjects will be asked to wear a measurement system (Eyelink II, SR Research) that tracks head and eye movements as they perform as set of eye and head movements to measure saccadic eye movements, VOR and VOR suppression. Periodic calibrations will be performed throughout the experiment to test the continued reliability of the data.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-04-18 (Actual); Study Completion 2017-04-18 (Actual)

PRIMARY OUTCOMES:
vestibulo-ocular reflex (VOR) gain | 2 hour data collection period (Visit 1)
  amplitude of head v. eye velocities
NASA Task Load Index | Immediately after 2 hour data collection period (Visit 1)
  measure of cognitive load during task performance

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pidcoe, PT, DPT, Ph.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No